CLINICAL TRIAL: NCT01022489
Title: Evaluation of Repetitive Transcranial Magnetic Stimulation (rTMS) at High Frequency With Neuronavigation in the Treatment of Auditory Hallucinations : A Randomized Multicentric Controlled Study
Brief Title: High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in Schizophrenia : a Randomized Controlled Study
Acronym: TMS-Hz
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-A01589-46
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Auditory Hallucinations in Patients With Schizophrenic Disorders
Keywords: Schizophrenia, auditory hallucinations, TMS
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial magnetic stimulation: rTMS (Experimental): rTMS : 4 sessions of 13 minutes, with 2 sessions a day, at 20Hz frequency and at an intensity of 80% of rest motor threshold will be delivered
  Interventions: Device: Transcranial magnetic stimulation: rTMS
- placebo (sham coil) treatment (Placebo Comparator)
  Interventions: Device: Placebo (sham coil) treatment

INTERVENTIONS:
Device: Transcranial magnetic stimulation: rTMS — 4 sessions of 13 minutes, with 2 sessions a day, at 20Hz frequency and at an intensity of 80% of rest motor threshold will be delivered
  Arms: Transcranial magnetic stimulation: rTMS
Device: Placebo (sham coil) treatment — Sham coil treatment
  Arms: placebo (sham coil) treatment

SUMMARY:
Background:

Repetitive transcranial magnetic stimulation (rTMS) is a recent therapeutic which has demonstrated its efficacy in the treatment of auditory hallucinations in patients with schizophrenic disorders. Up to now, the target of stimulation has been over the left temporoparietal region (based on the international 10-20 EEG system) and rTMS has been delivered at low frequency (1 Hz).

High frequency (20 Hz) might allow shortening the duration of treatment and so could be more convenient for the patient (2 days at high frequency instead of 15 days at low frequency).

Besides high frequency, an accurate target taking into account the inter-subjects anatomical variability might increase the efficacy. Based on a great overlap of language and auditory hallucinations networks, the investigators hypothesized that targeting the stimulation on the highest cluster of activation induced by a language task could be an easier and relevant method to determine the target. The investigators suggest that the best area is located at the posterior part of the left superior temporal sulcus (STS). Indeed, this area is considered as an " epicenter " of language, i.e., involved both in understanding and production of language and in the auditory hallucination network. Therefore, the investigators conducted an open pilot study in order to test the interest of rTMS at high frequency (20 Hz) associated with anatomical and functional magnetic resonance imaging (MRI) and neuronavigation in 11 schizophrenic patients with hallucinations. The investigators showed a significant reduction of auditory hallucinations; Seven out of 11 patients (63.8%) were considered as responders at day 12 with a decrease of more than 30% of the score of Hoffman's scale (Auditory Hallucinations Rating Scale) ; 2 patients presented a drastic improvement with no hallucinations after 12 days of rTMS. The investigators also showed the target based on anatomical and functional MRI was located at the intersection of the left STS and the coronal slice across the vertical line of sylvius sulcus.

The aim of this multicentric double-blind study (randomized and placebo sham) is to demonstrate the efficacy of rTMS at high frequency with neuronavigation in the treatment of auditory hallucinations in patients with schizophrenia and schizo-affective disorders (DSMIV-R).

Methods:

72 subjects will be included after written consent. After randomization, the subject will receive in a double blind either active treatment or placebo (sham coil) treatment.

rTMS : 4 sessions of 13 minutes, with 2 sessions a day, at 20Hz frequency and at an intensity of 80% of rest motor threshold will be delivered. These parameters allow the investigators to be under the risk of epilepsia, the only one severe side effect. Another mild side effect is headache easily treated by antalgic drugs. The target will be established with anatomical MRI eventually associated with functional MRI before treatment.

The efficacy of treatment will be evaluated over 4 weeks (D0, D1, D2, D7, D14, D21 and D30). The primary assessment is the percentage of patients who present a decrease of more than 30% of the frequency item of Auditory Hallucinations Rating Scale (AHRS) between D1 and D30 at 2 evaluations spaced of 1 week (Responder patients). The secondary assessments are : 1- Relative decrease of frequency item of AHRS between D1 and D14 ; 2- Evolution of total score of AHRS at D1, D2, D7, D14, D21 and D30 ; 3- Variation of scores of CGI, SUMD, IS, positive, negative, general and total PANSS scores between D0 and D14 and D30 ; 4- Scores at secondary side effects (adapted UKU) at D2 and D7; 5- Distances between the present target and the classical target based on 10-20 EEG system (T3P3) and/or the target established with functional MRI (cluster of activations induced by a listening comprehension task).

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenic disorders aged from 16 to 65 years old
* Patients suffering from auditory hallucinations (score AHRS > 10) undergoing antipsychotic treatments
* patients clinically stabilised (no antipsychotic treatments modifications for the last 2 months
* Written signed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* patients with a brain tumor
* Patients with previous history of epilepsy
* Patients already treated once by rTMS
* Counter-indication to MRI or to rTMS

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary assessment is the percentage of patients who present a decrease of more than 30% of the frequency item of AHRS between D1 and D30 at 2 evaluations spaced of 1 week (Responder patients) | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Dollfus, MD, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France